CLINICAL TRIAL: NCT04154345
Title: Exercise Into Pain in Chronic Rotator Cuff Related Shoulder Pain: a Prospective Single-Group Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University of Malaga (Other); Rotterdam University of Applied Sciences (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Filip Struyf, Professor, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/34/379
Record Dates: First submitted 2019-10-25; First posted 2019-11-06 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Prospective single-group study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Painful exercises (Experimental): The pain allowed during exercises ranges between 4 and 7 on NPRS (Numeric Pain Rating Scale)
  Interventions: Other: Exercise therapy (exercising into pain)

INTERVENTIONS:
Other: Exercise therapy (exercising into pain) — The intervention consists of 12 weeks of progressive loaded exercises, three times per week. There are 9 sessions of supervised physiotherapy treatment, lasting 30 minutes, while the rest of the sessions is conducted as home exercises. There are 4 strengthening exercises, in which the pain allowed ranges between 4 and 7 on a verbal NPRS for 9 weeks, then pain ratings are 0-2 for the remaining 3 weeks. Every physiotherapy session includes also 15 minutes of manual therapy.

SUMMARY:
The purpose of this study is to evaluate a) the feasibility of applying a painful exercise program in the treatment of subacromial shoulder pain and b) the time needed to collect clinical outcomes for a future randomized controlled trial.

DETAILED DESCRIPTION:
Exercise therapy is the first choice of treatment in the management of subacromial shoulder pain (SSP). Guidelines suggest active rehabilitation program for at least three months and existing research highlights the importance of progressive loaded exercise therapy at higher dosage. However, it is not clear which is the best type of exercise and if pain should be provoked during exercise. Recent research found that painful exercises are beneficial in short term on pain and function in patients with different kinds of chronic musculoskeletal pain. The aim of the future randomized clinical trial is to investigate if "exercising into pain" gives better results in term of clinical outcomes compared to a non-painful exercise program. Since the intervention consists in painful exercises, it is essential to test the rate of adherence in the intervention group (both during physiotherapist-led session and home-based exercises). Moreover, the practicability of clinical questionnaire via online survey will be tested and the time needed to collect clinical data will be calculated as well. Furthermore, feedback from physiotherapists and participants will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Shoulder pain for at least 3 months
* Pain in the antero-lateral shoulder region
* At least 3 out of 5 of the following tests positive: Neer test, Hawkins-Kennedy, Jobe, painful arc between 60° and 120°, external resistance test
* Resting pain should be at 2/10 maximum on verbal NRS scale
* All types of occupations were included: students, workers (including overhead workers or heavy duty workers), people on sick leave and retired people

Exclusion Criteria:

* Bilateral shoulder pain
* Corticosteroid injections 6 weeks prior to the study
* Pregnancy, inability to understand spoken or written Dutch
* Clinical signs of full-thickness rotator cuff tears (positive external and internal rotation lag tests and drop arm test)
* Evidence of adhesive capsulitis (50% or more than 30° loss of passive external rotation)
* Previous cervical, thoracic or shoulder surgery; recent fractures or dislocations on the painful shoulder
* Symptoms of cervical radiculopathy as primary complaint (tingling, radiating pain in the arm associated with neck complaints)
* Primary diagnosis of acromioclavicular pathology, shoulder instability
* A radiologically confirmed fracture or presence of calcification larger than 5 mm
* Presence of competing pathologies (inflammatory arthritis, neurological disorders, fibromyalgia, malignancy)
* More than 4h of training in sport overhead shoulder activities per week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Struyf, Professor, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Physiotherapy private practices, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cavaggion C, Juul-Kristensen B, Luque-Suarez A, Voogt L, Wollants G, O Conaire E, Struyf F. Exercise into pain in chronic rotator cuff related shoulder pain: a prospective single-group feasibility study. BMJ Open. 2023 Oct 6;13(10):e070698. doi: 10.1136/bmjopen-2022-070698. PMID 37802620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Painful Exercises
Started | 12
Completed | 8
Not Completed | 4
Not completed — Covid-19 pandemic | 4

BASELINE CHARACTERISTICS:
Arm/Group | Painful Exercises
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.5 [37 to 53.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 23.2 [21.3 to 24.8]
duration of symptoms [Median (Inter-Quartile Range); unit: months] | 6.5 [4 to 15.3]
dominant side affected [Count of Participants; unit: Participants] | 7
previous treatment [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adherence (Physiotherapy Session)
Description: It is analysed in terms of attendance to the physiotherapist-led sessions. Good level of adherence is defined by attendance of 7/9 (78%) of physiotherapist led-sessions
Time Frame: measurement every session, final measure at the end of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Rate of Adherence (Adherence Home Exercises)
Description: It is analysed in terms of adherence to home exercises. Good level of adherence is achieved when patients completed at least 22 of 27 (81%) sessions. One session of non-supervised (home) exercise was considered completed when at least 80% of the total amount of sets and repetitions were executed as prescribed by the physiotherapist.
Time Frame: measurement every home exercise session, final measure at the end of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
Participants | 4

3. Primary Outcome: Shoulder Pain and Disability Index (SPADI)
Description: There are 13 items, divided in two subscales: pain (5 items) and function (8 items). Each item is scored from 0 (no pain/no difficulty) to 10 (worst imaginable pain/so difficult it requires help) on a NPRS. The final score is a percentage derived from an average of the two subscales, where higher score means worse outcome.
Time Frame: value at baseline minus value at 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
score on a scale | 29.3 [13.8 to 75.9]

4. Secondary Outcome: Fear-Avoidance Beliefs Questionnaire (FABQ-PA)
Description: Fear-Avoidance Beliefs Questionnaire, Subscale Physical Activity (range: 0-24) Higher scores indicate higher fear-avoidance beliefs
Time Frame: value at baseline minus value at 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
score on a scale | 1.5 [-3 to 18]

5. Secondary Outcome: Fear-Avoidance Beliefs Questionnaire (FABQ-W)
Description: Fear-Avoidance Beliefs Questionnaire, Subscale Work (range: 0-42) Higher scores indicate higher fear-avoidance beliefs
Time Frame: value at baseline minus value at 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
score on a scale | 3 [-18 to 16]

6. Secondary Outcome: Fear of Pain Questionnaire (FPQ-9)
Description: It is a shortened version of the Fear of Pain Questionnaire-III. The total score ranges between 9 and 45.
  Higher scores indicate more fear and anxiety associated with pain.
Time Frame: value at baseline minus value at 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
score on a scale | 0 [-6 to 17]

7. Secondary Outcome: Passive Range of Motion (ROM) in External Rotation
Description: It is measured with the inclinometer. The unit of measure is degrees. Higher values indicate higher ROM.
Time Frame: value at 12 weeks minus baseline
Population: Data on passive ROM in external rotation were lost for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: degrees
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
degrees | 4 [-21 to 22]

8. Secondary Outcome: Passive ROM in Internal Rotation
Description: It is measured with the inclinometer. The unit of measure is degrees. Higher values indicate higher ROM.
Time Frame: value at 12 weeks minus baseline
Population: Data on passive ROM in internal rotation were lost for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: degrees
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
degrees | 1 [-21 to 22]

9. Secondary Outcome: Passive ROM in Scaption
Description: It is measured with the inclinometer. The unit of measure is degrees. Higher values indicate higher ROM.
Time Frame: value at 12 weeks minus baseline
Population: Data on passive ROM in scaption were lost for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: degrees
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
degrees | 27 [11 to 49]

10. Secondary Outcome: Active ROM in External Rotation
Description: It is measured with the inclinometer. The unit of measure is degrees. Higher values indicate higher ROM.
Time Frame: value at 12 weeks minus baseline
Population: Data on active ROM in external rotation were lost for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: degrees
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
degrees | 6 [-32 to 22]

11. Secondary Outcome: Active ROM in Internal Rotation
Description: It is measured with the inclinometer. The unit of measure is degrees. Higher values indicate higher ROM.
Time Frame: value at 12 weeks minus baseline
Population: Data on active ROM in internal rotation were lost for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: degrees
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
degrees | -4 [-38 to 8]

12. Secondary Outcome: Active ROM in Scaption
Description: It is measured with the inclinometer. The unit of measure is degrees. Higher values indicate higher ROM.
Time Frame: value at 12 weeks minus baseline
Population: Data on active ROM in scaption were lost for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: degrees
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
degrees | 24 [7 to 43]

13. Secondary Outcome: Maximum Voluntary Contraction (MVC) in External Rotation
Description: It is measured with the hand-held dynamometer. The unit of measure is Newtons. Higher values indicate greater strength.
Time Frame: value at 12 weeks minus value at baseline
Population: Data on MVC in external rotation were not collected at 12 weeks for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is not possible to present change between baseline and 12 weeks for 6 patients.
Measure: Median (Full Range); unit: Newtons
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
Newtons | 14.55 [-44.79 to 30.40]

14. Secondary Outcome: MVC in Internal Rotation
Description: It is measured with the hand-held dynamometer. The unit of measure is Newtons. Higher values indicate greater strength.
Time Frame: values at 12 weeks minus values at baseline
Population: Data on MVC in internal rotation were not collected at 12 weeks for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is not possible to present change between baseline and 12 weeks for 6 patients.
Measure: Median (Full Range); unit: Newtons
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
Newtons | 26.64 [-25.50 to 34.98]

15. Secondary Outcome: MVC in Scaption
Description: It is measured with the hand-held dynamometer. The unit of measure is Newtons. Higher values indicate greater strength.
Time Frame: values at 12 weeks minus baseline
Population: Data on MVC in scaption were not collected at 12 weeks for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients), while one value was lost because of an error during the measurement process. Therefore, it is possible to present change between baseline and 12 weeks only for 5 patients.
Measure: Median (Full Range); unit: Newtons
Arm/Group | Painful Exercises
Number analyzed (Participants) | 5
Newtons | 6.54 [-40.54 to 30.07]

16. Other Pre Specified Outcome: Acromiohumeral Distance (AHD)
Description: It is measured with the Ultrasound machine at rest and at 60 degrees of elevation in the scapular plane. (in millimeters)
Time Frame: value at baseline minus value at 12 weeks
Population: Data on ultrasonographic measures were not collected at 12 weeks for 6 out of 12 patients because of reasons related to COVID-19 (restrictions and/or illness of the patients). Therefore, it is possible to present change between baseline and 12 weeks only for 6 patients.
Measure: Median (Full Range); unit: millimeters
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
millimeters | 0.00 [-1.48 to 1.13]

17. Other Pre Specified Outcome: Supraspinatus Tendon Thickness (STT)
Description: It is measured with the Ultrasound machine in the Crass position (in millimeters)
Time Frame: value at baseline minus value at 12 weeks
Population: as for outcome 16
Measure: Median (Full Range); unit: millimeters
Arm/Group | Painful Exercises
Number analyzed (Participants) | 6
millimeters | -0.17 [-0.95 to 0.72]

18. Other Pre Specified Outcome: Global Perceived Effect - Recovery (GPE-R)
Description: The Global Perceived Effect (GPE) of recovery was measured after 1 week of treatment, at 6 week and at 12 weeks with the question: "To what extent do you feel recovered compared to the beginning of the treatment?" (from 1=very much better to 7=very much worse). Higher scores indicate worse outcome.
Time Frame: value at baseline minus value at 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
score on a scale | 3 [-1 to 3]

19. Other Pre Specified Outcome: Global Perceived Effect - Satisfaction (GPE-S)
Description: The Global Perceived Effect (GPE) of satisfaction was measured after 1 week of treatment, at 6 week and at 12 weeks with the question "To what extend are you satisfied about your treatment?" (from 1=absolutely satisfied to 7=absolutely dissatisfied). Higher scores indicate worse outcome.
Time Frame: value at baseline minus value at 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Painful Exercises
Number analyzed (Participants) | 8
score on a scale | 1 [-1 to 1]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Description of other (non-serious) adverse effects monitored during the study: when patients were leaving the study because of treatment-related reasons.
Arm/Group | Painful Exercises
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Limitations of the feasibility study are specified in the published article

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04154345/Prot_SAP_000.pdf